CLINICAL TRIAL: NCT04529070
Title: Nightmare Rescripting and Rehearsal: Testing a 10-Minute Intervention to Treat Recurring Distressing Dreams in Primary Care.
Brief Title: Nightmare Rescripting and Rehearsal
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Funding and PI separated from the Air Force
Sponsor: David Moss (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, David Moss, Principal Investigator, Mike O'Callaghan Military Hospital
Organization: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FWH20200116H
Record Dates: First submitted 2020-08-21; First posted 2020-08-27 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Nightmare; Sleep
Keywords: nightmare rescripting; dreams; behavioral health; sleep
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention + Standard of care (Experimental): Nightmare Rescripting and Rehearsal: a 10 minute intervention for Primary Care plus Sleep Hygiene handout.
  Interventions: Behavioral: Nightmare Rescripting and Rehearsal; Behavioral: standard of care
- Standard of care (Active Comparator): Standard of Care Sleep Hygiene handout alone.
  Interventions: Behavioral: standard of care

INTERVENTIONS:
Behavioral: Nightmare Rescripting and Rehearsal — This study aims to test the efficacy of an abbreviated version of Imagery Rehearsal Therapy ('Nightmare Rescripting and Rehearsal Therapy' (NRRT)) administered by non-mental health professionals in a Primary Care setting.
  Arms: Intervention + Standard of care
Behavioral: standard of care — standard of care

SUMMARY:
This study aims to test the efficacy of an abbreviated version of Imagery Rehearsal Therapy administered by non-mental health professionals in a Primary Care setting. This treatment, to be called 'Nightmare Rescripting and Rehearsal Therapy' (NRRT) would arm Primary Care medical personnel with a nonpharmacologic, ten minute intervention for treating recurring nightmares.

The study will provide sleep hygiene education to both the control and experiment groups, NRRT to the experiment group only, and compare their Nightmare Distress Questionnaire and Nightmare Frequency Tool at two (2), four (4), and six (6) week intervals.

DETAILED DESCRIPTION:
This is a prospective Randomized Controlled Trial to determine if a standard of care sleep hygiene handout plus a brief 10 minute intervention for recurring nightmares (Nightmare Rescripting and Rehearsal Therapy) reduces scores on the Nightmare Distress Questionnaire and Nightmare Frequency Tool, when compared to patients solely receiving a handout outlining sleep hygiene techniques. Individuals with a minimum score on the Nightmare Distress Questionnaire and Nightmare Frequency Tool of 15 out of a possible 52 who meet all other inclusion criteria will be invited to participate.

A clinically significant reduction will be considered if a decrease in Nightmare Distress and Frequency measures is greater than or equal to 25% from baseline. Secondary outcomes will include PCL-5 (PTSD), PHQ9 (Depression), GAD7 (Anxiety), ISI (Insomnia Severity Index) scores.

ELIGIBILITY:
**Patients must be able to get care at Nellis Air Force Base (a military installation) in order to participate in this study**

Inclusion Criteria:

* Active Duty members and DoD beneficiaries.
* Aged 18 years or older
* Recurring disturbing dreams (at least three times per month for the past one month)
* Participants must score a 15 out of a possible 52 on the Nightmare Distress Questionnaire and Nightmare Frequency Tool in order to qualify.

Exclusion Criteria:

* Aged less than 18 years old
* Unwilling to refrain from taking an over the counter or prescription medication for the purpose of improving sleep during the course of the study.
* Participants that score less than a 15 out of a possible 52 on the Nightmare Distress Questionnaire and Nightmare Frequency will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
Nightmare distress Questionnaire (change from nightmare distress baseline from screening at each 4 visits) | screening, visit 1 (week 0), visit 2 (week 2 +/- 1 week), visit 3 (week 4 +/- 1 week), visit 4 (week 6 +/- 1 week)
  13 questions, 0-4. 0 indicates lower level of distress and effects as related to nightmares.
Nightmare Frequency in the past week (change from nightmare frequency screening baseline at each 4 visits) | screening, visit 1 (week 0), visit 2 (week 2 +/- 1 week), visit 3 (week 4 +/- 1 week), visit 4 (week 6 +/- 1 week)
  Boxes numbered one to 31. Pt circles the number corresponding to the number of days they had a nightmare in the past month.

SECONDARY OUTCOMES:
Posttraumatic Stress Disorder Checklist (PTSD) | screening, visit 1 (week 0), visit 2 (week 2 +/- 1 week), visit 3 (week 4 +/- 1 week), visit 4 (week 6 +/- 1 week)
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The questionnaire is self-report and may be completed in 5-10 minutes. Lower score indicates less severity of PTSD symptoms but is broad enough to pick up a wide base of patients with possible PTSD. Higher scores indicate greater severity and also offeres greater sensitivity.
Beck Depression Inventory II | screening, visit 1 (week 0), visit 2 (week 2 +/- 1 week), visit 3 (week 4 +/- 1 week), visit 4 (week 6 +/- 1 week)
  BDI-II. This questionnaire self-report and is made up of 21 groups of statements designed to measure attitudes and symptoms of depression severity. Each question has options that are scored on a scale of 0 to 3. Higher scores equals more severity of depression symptoms.
General Anxiety Disorder (anxiety) | screening, visit 1 (week 0), visit 2 (week 2 +/- 1 week), visit 3 (week 4 +/- 1 week), visit 4 (week 6 +/- 1 week)
  GAD-7. Objective screening tool to use to identify severity of: (Generalized Anxiety Disorder, Panic Disorder, Social Phobia and PostTraumatic Stress Disorder). 7 questions with options 0-3 and with a higher score indicating greater symptom severity.
Insomnia Severity Index (insomnia) | screening, visit 1 (week 0), visit 2 (week 2 +/- 1 week), visit 3 (week 4 +/- 1 week), visit 4 (week 6 +/- 1 week)
  ISI. Measures insomnia problems occurring in the last 2 weeks. 7 questions with added up scores. Higher score indicates greater symptom severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Mike O'Callaghan Military Medical Center, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing data.

REFERENCES:
- [Background] American Psychiatric Association. (2013). Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition. Arlington, VA: American Psychiatric Association.
- [Background] Belicki K. (1992). The relationship of nightmare frequency to nightmare suffering with implications for treatment and research. Dreaming 2 143-148. 10.1037/h0094355
- [Background] Böckermann, M., Gieselmann, A., & Pietrowsky, R. (2014). What does nightmare distress mean? Factorial structure and psychometric properties of the Nightmare Distress Questionnaire (NDQ). Dreaming, 24(4), 279-289. https://doi.org/10.1037/a0037749
- [Background] Collen JF, Williams SG, Lettieri CJ. Doomed to Repeat History: The Burden of Trauma-Related Nightmares in Military Personnel. J Clin Sleep Med. 2018 Mar 15;14(3):303-305. doi: 10.5664/jcsm.6964. No abstract available. PMID 29458710
- [Background] Creamer JL, Brock MS, Matsangas P, Motamedi V, Mysliwiec V. Nightmares in United States Military Personnel With Sleep Disturbances. J Clin Sleep Med. 2018 Mar 15;14(3):419-426. doi: 10.5664/jcsm.6990. PMID 29510796
- [Background] Harb, G. C., Forbes, D., Phelps, A., Gehrman, P. R., Cook, J. M., Gamble, G. & Ross, R. J. (2010). Treatment Manual for Imagery Rehearsal + cCBT for Insomnia.
- [Background] Köthe, M. & Pietrowsky, R. (2001). Behavioral effects of nightmares and their correlations to personality patterns. Dreaming, 11, 43-52.
- [Background] Krakow B, Kellner R, Neidhardt J, Pathak D, Lambert L. Imagery rehearsal treatment of chronic nightmares: with a thirty month follow-up. J Behav Ther Exp Psychiatry. 1993 Dec;24(4):325-30. doi: 10.1016/0005-7916(93)90057-4. PMID 8077451
- [Background] Krakow B, Hollifield M, Schrader R, Koss M, Tandberg D, Lauriello J, McBride L, Warner TD, Cheng D, Edmond T, Kellner R. A controlled study of imagery rehearsal for chronic nightmares in sexual assault survivors with PTSD: a preliminary report. J Trauma Stress. 2000 Oct;13(4):589-609. doi: 10.1023/A:1007854015481. PMID 11109233
- [Background] Levin R, Nielsen TA. Disturbed dreaming, posttraumatic stress disorder, and affect distress: a review and neurocognitive model. Psychol Bull. 2007 May;133(3):482-528. doi: 10.1037/0033-2909.133.3.482. PMID 17469988
- [Background] Pruiksma, K. E., Slavish, D., Wardle, S. Ojeda, A., Taylor, D., Peterson, A., Kelly, K., Maur, D., Mintz, J., Litz, B., Borah, E., Brundige, A., Young-McCaughan, S., Williamson, D. (2019). Prevalence and correlates of nightmares in Active Duty Service Members. Sleep, (42)1, A267. https://doi.org/10.1093/sleep/zsz067.667
- [Background] Seda G, Sanchez-Ortuno MM, Welsh CH, Halbower AC, Edinger JD. Comparative meta-analysis of prazosin and imagery rehearsal therapy for nightmare frequency, sleep quality, and posttraumatic stress. J Clin Sleep Med. 2015 Jan 15;11(1):11-22. doi: 10.5664/jcsm.4354. PMID 25325592